CLINICAL TRIAL: NCT05017818
Title: A Retrospective Study of Subjects With Thymidine Kinase 2 Deficiency Treated With the Combination of Pyrimidine Nucleos(t)Ides as Well as Untreated Subjects to Collect Vital Status Data and Supporting Information
Brief Title: A Retrospective Study of Subjects With Thymidine Kinase 2 Deficiency
Status: Completed | Type: Observational
Sponsor: Zogenix MDS, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: MT-1621-107
Record Dates: First submitted 2021-07-12; First posted 2021-08-24 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Thymidine Kinase 2 Deficiency
Keywords: TK2D; mitochondrial disorder; mitochondrial disease; mitochondria; primary mitochondrial myopathy; mitochondrial depletion syndrome; muscle weakness; muscle atrophy; loss of mobility
MeSH Terms: conditions — Mitochondrial Diseases; Muscle Weakness; Muscular Atrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treated and untreated subjects with TK2 deficiency: Two TK2 deficiency groups. (1) Subjects treated with chemical-grade dCMP/dTMP, dC/dT, and/or MT1621 outside of a Modis sponsored study. (2) Subjects not treated with chemical-grade dCMP/dTMP, dC/dT, and/or MT1621 outside of a Modis sponsored study.
  Interventions: Other: Observational retrospective data

INTERVENTIONS:
Other: Observational retrospective data — Non-intervention

SUMMARY:
This is a multicenter, multinational, retrospective chart-review study to evaluate survival in patients with Thymidine Kinase 2 deficiency (TK2d).

DETAILED DESCRIPTION:
This is a retrospective, chart-review study. The primary goal is to use data on survival and other related information to support a comprehensive evaluation of patients with Thymidine Kinase 2 deficiency (TK2d) who have not been treated with pyrimidine nucleos(t)ides including deoxycytidine monophosphate/deoxythymidine monophosphase (dCMP/dTMP), and deoxycytidine/deoxythymidine (dC/dT), and/or MT1621(dC/dT), and those that have received one or more of these treatments. The secondary goals of this study will focus on describing the participant's clinical course and treatment experience.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the subject or parent(s)/LAR and/or assent by the subject (when applicable), unless the associated IRB or EC provides an appropriate consent waiver that allows review of medical records for this study.
2. Confirmed genetic mutations in the TK2 gene.
3. Availability of medical records or information pertaining to vital status at a minimum.

Exclusion Criteria:

Not applicable as this is a non-interventional study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Thymidine Kinase 2 deficiency
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Number of participants who have died. | Start of observation period (first medical record available on site), to last medical record available on site or end of observation period on 12-Jan-2022, whichever comes first.
  Participant date of death or date last known alive.

SECONDARY OUTCOMES:
Change from baseline in development motor milestones. | Start of observation period (first medical record available on site), to last medical record available on site or end of observation period on 12-Jan-2022, whichever comes first.
  Modified motor milestones as defined by World Health Organization include: Ability to Hold head upright, unassisted; Ability to roll from supine to sides; Ability to sit upright, unassisted; Ability to sit upright, slightly assisted; Ability to raise self and stand; Ability to stand, unassisted; Ability to stand, assisted; Ability to walk, unassisted; Ability to walk, assisted; Ability to climb stairs, unassisted; Ability to climb stairs, assisted; Ability to jump; Ability to hop; Ability to run
Change from baseline in feeding support. | Start of observation period (first medical record available on site), to last medical record available on site or end of observation period on 12-Jan-2022, whichever comes first.
  Feeding support includes gastrostomy tube or nasogastric tube.
Change from baseline in respiratory support. | Start of observation period (first medical record available on site), to last medical record available on site or end of observation period on 12-Jan-2022, whichever comes first.
  Respiratory support includes non-invasive ventilation (e.g. bi-level positive airway pressure [Bi-PAP]) and mechanical ventilation.
Clinical Global Impression of Improvement (CGI-I). | Start of observation period (first medical record available on site), to last medical record available on site or end of observation period on 12-Jan-2022, whichever comes first.
  The CGI-I is a 7-point Likert scale would have been conducted by a physician or trained rater at a clinic visit to establish overall clinical change.
Number of participants with treatment-emergent adverse events (AEs) or serious adverse events (SAEs) that cause a decrease in dose or a stop in dosing (temporary or permanent). | Start of observation period (first medical record available on site), to last medical record available on site or end of observation period on 12-Jan-2022, whichever comes first.
  An AE is any untoward medical occurrence in a participant that was receiving treatment without regard to causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly. SAEs were AEs excluding non-serious AEs.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, MD, Study Director — 001 844 599 2273
Locations (12):
- United States (4):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Akron Children's Hospital, Akron, Ohio
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
- Russia (2):
  - Medical Center Zdorovyy Rebenok, Voronezh, Voronezh Oblast
  - NIKI Pediatrii im Veltischeva, Children's Neuromuscular center, Moscow
- Spain (4):
  - Vall d'Hebron Institut de Recerca, Barcelona
  - Hospital Clínic Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Turkey (Türkiye) (2):
  - Istanbul Universitesi, Istanbul Tip Fakultesi, Fatih, Istanbul
  - Yeditepe University Koşuyolu Hospital, Kadiköy